CLINICAL TRIAL: NCT05398172
Title: Clinical Evaluation of Fractional Bi-Polar Radio-Frequency for Symptoms of Vulvovaginal Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO610363A
Record Dates: First submitted 2022-05-17; First posted 2022-05-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Vaginal Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- treatment (Experimental): 3 treatments once a month
  Interventions: Device: MorpheusV Applicator

INTERVENTIONS:
Device: MorpheusV Applicator — Eligible subjects will receive 3 treatments 4 weeks apart with the MorpheusV Applicator according to the study protocol

SUMMARY:
Prospective, one arm, baseline-controlled At least 30 healthy adult female volunteers, from 2 investigational sites seeking treatment for Symptoms of Vulvovaginal Atrophy Eligible subjects will receive 3 treatments 4 weeks apart with the MorpheusV Applicator according to the study protocol The subject will return for 3 follow up visits: 3 months follow up (3M FU), 6 months follow up (6M FU), 12months follow up (12M FU) after the treatment.

Total expected study duration is approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study.
* BMI < 36
* VHIS<15
* Healthy non-smoking female subjects, > 35 and < 75 years of age at the time of enrolment post menopausal with absence of menstruation of at least 12 months
* General good health confirmed by medical history and examination of the treated area.
* The patients should be willing to comply with the study procedure and schedule, including the follow up visit, and will refrain from using any other treatment methods in the treated area for the last 6 months and during the entire study period.

Exclusion Criteria:

* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
* Permanent implant in the treated area such as metal plates and screws, silicone implants or an injected chemical substance, unless deep enough in the periostal plane.
* Current or history of skin cancer, or current condition of any other type of cancer, or premalignant moles.
* Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Pregnancy and nursing.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* History of bleeding coagulopathies or use of anticoagulants in the last 10 days.
* Any surgery in treated area within 3 months prior to treatment.
* Simultaneous participation in another investigator drug or device study or completion of the follow-up phase for the primary endpoint of any previous study less than 30 days prior to the first evaluation in this study.
* Six months delay is required if other recent treatments like light, CO2 laser or RF were performed on the same area.
* Acute urinary tract infection (UTI), or genital infection (e.g. IVU, herpes genitalis, candida).
* Treatment with any Vaginal Estrogen medication within 30 days
* Prolapse beyond hymen
* Any chronic condition that could interfere with study compliance
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the patient

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
effect of treatment on VVA symptoms, | baseline through 12 months
  effect of treatment on VVA symptoms, such as pain, vaginal burning, vaginal itching, dyspareunia and dysuria, using the Visual Analog Scale (VAS). scored from 1 to 10, the lower the score the better the outcome
objective evaluation of vaginal atrophy/estrogenization | baseline through 12 months
  measured by the globally validated "Vaginal Health Index" (VHI) score at follow up visits 3M, 6M FU and 12M FU) compared to Baseline. Scored from 5 to 25, the higher the score the better the outcome
Assess the effect of treatment on the general quality of life, | baseline through 12 months
  by mean of the "Short Form 12" (SF-12) specific questionnaire. Administered at baseline and at follow up visits 3M, 6M and 12M FU).
The effect of the treatment on Sexual Function | baseline through 12 months
  measured by Female Sexual Function Index (FSFI) at follow up visits (3M FU,6M FU and 12M FU) compared to baseline. the higher the score the better the outcome
Assess the degree of difficulty encountered by the physician in performing the treatment, | baseline through 12 months
  by mean of a 5-point Likert scale. the higher the score the better the outcome
The rate of satisfaction of patients with treatment | baseline through 12 months
  assessed by the Patient Global Impression of Improvement (PGI), using a 5-point Likert scale. The subjects will answer this questionnaire at follow up visits 3M FU, 6M and 12M FU). the higher the score the better the outcome
The effect of the treatment on urinary symptoms | baseline through 12 months
  by means of Urogenital Distress Inventory 6 Questionnaire. Administered at baseline and at each follow up visit (3M FU, 6M FU, 12M FU). the lower the score the better the outcome

SECONDARY OUTCOMES:
Occurrence of expected post-treatment adverse events | up to 12 months
  Occurrence of expected post treatment immediate response including erythema and edema and during all study period based on predefined scale
Discomfort scale | up to 3 months
  A 10cm visual analog scale from 0 (no discomfort) to 10 (worst possible discomfort) to measure discomfort associated with probe insertion, and RF energy application at the treatment visit
Adverse events | baseline through 12 months
  Number, severity and type of any adverse event recorded throughout the course of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Beyond Regenerative Medicine and Aesthetics, Newport Beach, California
  - Institute for Female Pelvic Medicine, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided